CLINICAL TRIAL: NCT03739307
Title: Characterization & Treatment of Chronic Pain After Moderate to Severe Traumatic Brain Injury
Brief Title: Characterization & Treatment of Chronic Pain After Moderate to Severe TBI
Status: Completed | Type: Observational
Sponsor: Craig Hospital (Other)
Collaborators: University of Washington (Other); James A. Haley Veterans Administration Hospital (U.S. Federal Agency); Rehabilitation Hospital of Indiana (Other); Spaulding Rehabilitation Hospital (Other); Wayne State University (Other); Mayo Clinic (Other); Baylor Institute for Rehabilitation (Other); Virginia Commonwealth University (Other); NYU Langone Health (Other); University of Alabama at Birmingham (Other); Moss Rehabilitation Research Institute (Other); TIRR Memorial Hermann (Other)
Responsible Party: Principal Investigator, Cynthia Harrison-Felix, PhD, Co-Principal Investigator, Craig Hospital
Other Study IDs: 90DPTB0017-01-00
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Traumatic Brain Injury; Pain
MeSH Terms: conditions — Brain Injuries, Traumatic; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a five year multi-site, cross sectional, observational study designed to examine chronic pain and pain treatment after moderate to severe TBI.

DETAILED DESCRIPTION:
The aims of this study are to: 1) Determine chronic pain classification (musculoskeletal, headache, central/neuropathic), prevalence, location, duration, and associations with demographic, injury severity, current level of functioning and comorbidities in participants followed in ten Centers participating in the National Institute on Disability, Independent Living and Rehabilitation Research and the Department of Veterans Affairs TBIMS Databases; 2) Identify extreme groups based on responses to pain (interference and perception of improvement with treatment), or chronic pain extreme phenotypes, in order to define the key differences between those who have a good outcome and those who do not, across factors related to injury, pain severity/location, demographics, and treatment history; and 3) Identify treatment practices by clinicians who treat comorbid TBI and chronic pain to determine gaps in availability/accessibility of guideline level treatment, highlighting underserved populations where applicable.

Results from this study will provide a more detailed picture of the problem of chronic pain after TBI by examining the types of pain that occur after TBI, which may be multiple types of pain for a subset of individuals, as well as the frequency of comorbid conditions. Identifying extreme phenotypes, such as demographic, individual, and treatment factors associated with those who have chronic pain but have minimal interference compared to those who are significantly impacted by pain, will allow us to identify treatment targets (behavioral, cognitive, biological, and molecular) to advance a personalized medicine approach to treatment unlike any approach in TBI and chronic pain to date. Outcomes from this study will include educational materials on chronic pain and pain treatment to benefit patients, family members, clinicians, and policymakers. Data from this study will have a direct impact on clinical practice, informing future work, and promoting understanding of constituent factors in extreme phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled in the TBI Model Systems National Database (TBNIMS NDB) at one of the collaborating sites and thus will meet the TBIMS NDB criteria which are: (1) medical documentation of TBI caused by external mechanical force with either loss of consciousness exceeding 30 minutes, post-traumatic amnesia lasting more than 24 hours, Glasgow Coma Scale score in ER of less than 13, or trauma related intracranial abnormality or neuroimaging abnormalities; (2) admitted to the TBI inpatient rehab program at study sites; and (3) minimum age of 16 [18 for VA site]

Exclusion Criteria:

* Participants unable to participate in the surveys themselves will not be included (i.e. no proxy surveys).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants have sustained a moderate to severe TBI and are now being followed at the collaborating centers as part of the TBIMS NDB which is a study collecting observational data after TBI.
Sampling Method: Non-Probability Sample
Enrollment: 3805 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Each participant will complete assessment one time during 4 years of data collection
  The BPI will be used to determine pain intensity as well as interference related to pain. Intensity of pain is rated by participant on a scale of 0 (no pain) to 10 (pain as bad as you can imagine) when the pain is at it's "worst," "least," "average," and "right now." Pain interference is assessed with seven items using a numeric rating scale ranging from 0 (no interference) to 10 (complete interference). Participants are asked to rate how much pain has interfered with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life
painDetect Questionnaire | Each participant will complete assessment one time during 4 years of data collection
  This self report survey consists of seven questions about location and quality of neuropathic pain. Scores range from 0-38 with scores above 18 indicating neuropathic pain and higher scores indicating more severity of pain.

SECONDARY OUTCOMES:
Post-Traumatic Stress Disorder Checklist-5 (PCL-5) | Each participant will complete assessment one time during 4 years of data collection
  The PCL-5 is a 20-item, self-rating scale that provides a quick and accurate measure of PTSD symptoms. Responses are scored on Likert scale (0 = "Not at All" to 4 = "Extremely"). Total score of 0 to 80 with higher scores indicating more PTSD symptomatology
Pain Self Efficacy Questionnaire-2 (PSEQ-2) | Each participant will complete assessment one time during 4 years of data collection
  PSEQ-2 is designed to assess the level of confidence the respondent has in their ability to accomplish daily activities despite their pain. items are rated on a 7-point scale (0 = not at all confident to 6 = completely confident).
Coping Strategies Questionnaire (CSQ) | Each participant will complete assessment one time during 4 years of data collection
  An abbreviated version of the CSQ will be used to reduce patient burden. This version uses only two items per domain to assess four coping strategies associated with adjustment to chronic pain: catastrophizing, ignoring pain sensations, increasing behavior, and using coping self-statements. Each item is scored from 0 to 6, with 0 representing 'no use' and 6 representing 'regular use' of the coping strategy. Scores for each domain are the mean score of the two items in that domain.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama, Birmingham, Alabama
  - Craig Hospital, Englewood, Colorado
  - Tampa VA, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - Spaulding Rehabilitation Institute, Charlestown, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York University School of Medicine, New York, New York
  - MOSS Rehabilitation Research Institute, Elkins Park, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - TIRR Memorial Hermann, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington